CLINICAL TRIAL: NCT07225049
Title: Pilot of an Integrated Treatment for Comorbid PTSD and Chronic Pain
Brief Title: Integrated PTSD and Chronic Pain Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-01028464
Record Dates: First submitted 2025-10-27; First posted 2025-11-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: PTSD; Chronic Pain
Keywords: PTSD; Chronic Pain; Integrated Treatment; Comorbidity; Prolonged Exposure; CBT for Chronic Pain; Cognitive Behavioral Therapy for Chronic Pain
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrated PTSD and Chronic Pain Treatment (Experimental): Integrated treatment combining modules from Prolonged Exposure Therapy with Cognitive Behavioral Therapy for Chronic Pain
  Interventions: Behavioral: Integrated Treatment for PTSD and Chronic Pain

INTERVENTIONS:
Behavioral: Integrated Treatment for PTSD and Chronic Pain — The intervention consists of 12 90-minute virtual psychotherapy sessions scheduled twice per week. The treatment integrates modules from Prolonged Exposure and Cognitive Behavioral Therapy for Chronic Pain.

SUMMARY:
Posttraumatic stress disorder (PTSD) occurs in approximately 7% of adults in the general population. PTSD greatly impacts quality of life and often co-occurs with other conditions such as chronic pain. Individuals with co-morbid PTSD and chronic pain demonstrate higher PTSD symptoms and pain (as well as greater anxiety, depression, disability, and opioid use) compared to those with only one of those conditions. Gold standard treatments exist for both PTSD (e.g., Prolonged Exposure; PE) and chronic pain (e.g., Cognitive Behavioral Therapy for Chronic Pain; CBT-CP) and are generally offered sequentially (i.e., one at a time for the condition that is most prominent). Treating these conditions separately may overlook their interconnected nature, which may reduce efficacy and increase dropout. Thus, there is a need for an intervention to target both simultaneously, which may be more effective and efficient than treating conditions sequentially.

This is a single-arm pilot study to assess the feasibility and acceptability of an integrated treatment for adults with comorbid PTSD and chronic pain. The intervention consists of 12 90-minute virtual psychotherapy sessions scheduled twice per week. The treatment draws from modules in PE and CBT-CP including psychoeducation, exposure to feared/avoided situations and activities, processing of exposures, behavioral activation, breathing and relaxation techniques, sleep hygiene, symptom monitoring, and structured homework assignments. Baseline and post-treatment assessments will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English-speaking
* Currently meets criteria for PTSD, assessed by the CAPS-5 (any trauma type) - Chronic pain, assessed by greater than or equal to 4 on a scale of 0-10 pain severity over the past 3 months
* Medically stable at the time of study enrollment (chronic illness and disability does not prevent attendance of outpatient therapy sessions)
* Stable on psychotropic medication for past 60 days
* Agreed to not change current medication or pain-related treatments over the course of the study unless medically necessary

Exclusion Criteria:

* Lifetime diagnosis of schizophrenia, other psychotic disorder, or bipolar I disorder
* Participation in concurrent evidence-based psychological treatment for PTSD or chronic pain during the past 3 months
* Participants must not participate in an evidence-based psychological treatment for either PTSD or pain during the course of the study.
* Moderate or severe substance use in the past 90 days
* Cognitive impairment to the degree that the patient cannot provide informed consent or fill out assessment measures
* Participants who in the PI's judgement pose a current homicidal or suicidal risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility Indicator: Number of Participants Screened | Baseline
  Feasibility assessment will include number of participants screened defined as number of individuals who complete our initial eligibility screener.
Feasibility Indicator: Enrollment | Baseline
  Feasibility assessment will include enrollment defined as number of participants signing the informed consent form.
Feasibility Indicator: Number of Sessions Attended | Post-Treatment Assessment at approximately 6 weeks
  Feasibility assessment will include the number of sessions attended on average (out of 12).
Feasibility Indicator: Attrition Percentage | Post-Treatment Assessment at approximately 6 weeks
  A feasibility measure of attrition will be assessed by examining the percent of individuals who did not complete all 12 intervention sessions.
Feasibility Indicator: Number of Assessments Attended | Baseline and Post-Treatment Assessment at approximately 6 weeks
  A feasibility indicator of number of assessments (baseline and post-treatment) attended will be measured.
Feasibility Indicator: Percentage of Self-Reports Completed | Baseline, Post-Intervention at approximately 6 weeks, Every Other Treatment Session (Every 2 weeks up to 12 weeks)
  Self-reports are administered at each assessment (baseline and post-intervention) as well as every other treatment session (every 2 weeks up to 12 weeks). Therefore, there are 8 total self-report assessments and the percentage of those completed will be calculated.
Intervention Satisfaction | Post-Treatment Assessment at approximately 6 weeks
  Intervention satisfaction will be rated with a Likert scale ranging from 1-10 with greater scores indicating higher satisfaction.
Intervention Acceptability | Post-Treatment Assessment at approximately 6 weeks
  Intervention acceptability will be measured on a Likert scale ranging from 1-10 with greater scores indicating higher acceptability.
Qualitative Intervention Feedback | Post-Treatment Assessment at approximately 6 weeks
  Open-ended questions that include assessing overall impressions of treatment, feedback on the frequency and length of sessions, challenges or barriers, likelihood of recommending this treatment to a friend, and comparison of this treatment to other treatments received in the past.

SECONDARY OUTCOMES:
Change in Score on the Clinician Administered PTSD Score (CAPS-5) | Baseline to approximately 6 weeks
  Change in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Score. Total Scores range from 0-80. Higher scores indicate greater symptom severity.
Change in Score on the PTSD Checklist for DSM-5 (PCL-5) | Baseline to approximately 6 weeks
  The well-validated PCL-5 will assess self-reported PTSD symptom severity. Scores range from 0-80. Higher scores indicate greater symptom severity.
Change in Score on the Pain Severity Subscale of the Brief Pain Inventory (BPI) | Baseline to approximately 6 weeks
  Pain severity is a 4-item subscale with ranges from 0-10. Greater scores indicate higher pain severity.
Change in Score on the Pain Interference Subscale of the Brief Pain Inventory (BPI) | Baseline to approximately 6 weeks
  Pain interference is a 7-item subscale with ranges from 0-10. Greater scores indicate greater pain interference.
Change in Score on the Pain Catastrophizing Scale (PCS) | Baseline to approximately 6 weeks
  The 13-item PCS measure has scores ranging from 0-52, with higher scores indicating greater pain catastrophizing. Three subscales (rumination, magnification, and helplessness) are summed to form the total score.
Change in Score on the Chronic Pain Acceptance Questionnaire (CPAQ) | Baseline to approximately 6 weeks
  This 20-item measure results in a total score ranging from 0-120 with high scores reflecting greater acceptance of pain. Two subscales (activity engagement and pain willingness) are summed to create the total score.
Change in Score on the Posttraumatic Cognitions Inventory (PTCI) | Baseline to approximately 6 weeks
  The 33-item PTCI yields three subscores: negative cognitions about the self, negative cognitions about the world, and self-blame. Items are averaged so the range of scores for each subscale is 0-7 with higher scores representing more maladaptive cognitions. A total score is calculated by summing each of the 33 items yielding a score between 33-231, with higher scores indicating more maladaptive cognitions.
Change in Score on the Fear-Avoidance Components Scale (FACS) | Baseline to approximately 6 weeks
  This 20-item measure results in total scores ranging from 0-100, with greater scores indicating more severe fear-avoidance beliefs.
Change in Score on the Anxiety Sensitivity Index (ASI-3) | Baseline to approximately 6 weeks
  This 18-item measure results in a total score ranging from 0-72 with higher scores reflecting greater anxiety sensitivity. Three subscales (physical concerns, cognitive concerns, and social concerns) are summed to create a total score.
Change in Score on the Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST) | Baseline to approximately 6 weeks
  The ASSIST is a questionnaire that screens for all levels of problem or risky substance use in adults including tobacco, alcohol, cannabis, cocaine, amphetamine-type stimulants, inhalants, sedatives, hallucinogens, opioids, and other drugs. A score for each substance ranges from 0-39 with higher scores indicating greater problems or risks related to substance use. A total score is not computed and instead, each substance will be analyzed individually.
Change in Score on the Expectancies for Alcohol Analgesia (EAA) Measure | Baseline to approximately 6 weeks
  The EAA is a 5-item scale. Items are summed to generate a total score ranging from 0-45 with higher scores indicating greater expectancy for alcohol analgesia.
Change in Score on the Difficulties in Emotion Regulation Scale (DERS-18) | Baseline to approximately 6 weeks
  This 18-item measure results in a total score ranging from 18-90 with higher scores reflecting greater difficulties with emotion regulation.
Change in Score on the Patient Health Questionnaire (PHQ-9) | Baseline to approximately 6 weeks
  The PHQ-9 scores range from 0-27. Higher scores indicate greater symptom severity.
Change in Score on the Insomnia Severity Index (ISI) | Baseline to approximately 6 weeks
  7 item self-report measure. Total scores range from 0-28, with higher scores indicating higher insomnia severity.
Change in Score on the Multidimensional Assessment of Interoceptive Awareness (MAIA-2) | Baseline to approximately 6 weeks
  This is a 37-item measure that results in 8 subscales: noticing, not-distracting, not-worrying, attention regulation, emotional awareness, self-regulation, body listening, and trust. Each subscale ranges from 0-5, where higher scores reflect more awareness of bodily sensations. A total score is not computed, and instead, each subscale is analyzed individually.
Change in Score on the Quality of Life Inventory (QOLI) | Baseline to approximately 6 weeks
  The assessment yields an overall score and profile in 16 areas of life; health, self-esteem, goals and values, money, work, play, learning, creativity, helping, love, friends, children, relatives, home, neighborhood, and community. Subscales are computed by multiplying satisfaction (-3 to +3) by importance (0 to 2) and resulting scores are averaged to yield a total score ranging from -6 to +6, with higher scores indicate higher level of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn Difede, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No